CLINICAL TRIAL: NCT07230613
Title: Neo-adjuvant Intratumoral Anti-CTLA4 + Anti-PD1 in Patients With Localized Melanoma
Brief Title: Neo-adjuvant Immunotherapy in Patients With Localized Melanoma
Acronym: NEOREM-NEO-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-IMM-2510; 2025-522127-95-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-26; First posted 2025-11-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Melanoma, Stage III; Mucosal Melanoma
Keywords: Neo-adjuvant Immunotherapy; Localized Cancers; Intra-tumoral treatment; Melanoma; Immune-checkpoint blockade
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Solutions; Nivolumab

STUDY DESIGN:
Intervention Model Description: NEO-1 is an academic, non-comparative, non-randomized, multicenter Phase II clinical trial evaluating the effectiveness and safety of intratumoral injections of ipilimumab combined with nivolumab as a neoadjuvant treatment for patients with operable, localized stage III cutaneous or mucosal melanoma. Eligible patients in the NEOREM master protocol and its therapeutic sub-protocol i.e. NEO-1 trial will receive three injections of the ipilimumab and nivolumab combination, one injection every three weeks over six weeks prior to surgery. Surgery will take place between 6 and 8 weeks after the last intratumoral injection. If deemed necessary by the doctor, some patients may receive standard adjuvant treatment after surgery. Patient participation in the trial will not exceed 65 months from their selection into NEOREM and inclusion in NEO-1 including the treatment, surgery and post-surgery follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm immunotherapy with Ipilimumab and nivolumab intra-tumoral administration (Experimental): Patients will receive up to 3 doses of neo-adjuvant treatment with IT injections of ipilimumab (5mg/mL) & nivolumab (10mg/mL) at 3-week intervals (±3 days) for up to 6 weeks prior to surgery.
  Interventions: Drug: Ipilimumab (YervoyTM, 50 mg/10 mL solution); Drug: Nivolumab (OpdivoTM, 40 mg/4mL solution)

INTERVENTIONS:
Drug: Ipilimumab (YervoyTM, 50 mg/10 mL solution) — The 25 mg flat dose of the Ipilimumab will be administered by intra-tumoral injection. Injections will be performed under image guidance (the most adequate according to investigators preference). Ultrasound guidance will be privileged, as it is not using radiation. A maximum of 3 intratumoral procedures may occur with 3 weeks intervals prior to surgery.
Drug: Nivolumab (OpdivoTM, 40 mg/4mL solution) — The 30 mg flat dose of the Nivolumab will be administered by intra-tumoral injection. Injections will be performed under image guidance (the most adequate according to investigators preference). Ultrasound guidance will be privileged, as it is not using radiation. A maximum of 3 intratumoral procedures may occur with 3 weeks intervals prior to surgery.

SUMMARY:
The success of anti-PD-1 and anti-CTLA-4 therapies has initiated a paradigm shift in oncology, with drugs now targeting the immune system rather than cancer cells to stimulate the antitumor immune response. Intratumoral (IT) delivery of immunostimulating agents reduces the systemic toxicity associated with monoclonal antibodies (mAbs) targeting immune checkpoints. Notably, IT injections of immune checkpoint blockade (ICB) have been shown to induce immune-mediated tumor responses both at the injected site and at distant, non-injected tumor sites. While surgery has traditionally been the preferred treatment for stage III and IV melanoma patients, neoadjuvant therapy with anti-CTLA-4 and anti-PD-1 agents has shown promising efficacy.

In patients with localized melanoma, it is hypothesized that IT administration of ipilimumab (anti-CTLA-4 Ab) combined with nivolumab (anti-PD-1 Ab) will provide the most effective and safe treatment combination.

The NEO-1 study is a proof-of-concept clinical trial designed as a sub-protocol of NEOREM master protocol (NCT07262489) to validate the intratumoral immunotherapy approach, aiming to maximize the dose/efficacy ratio of combined ipilimumab and nivolumab treatment while minimizing systemic adverse events. This is an academic, open-label, multicentric, phase II clinical trial evaluating the efficacy and safety of intratumoral injections of ipilimumab and nivolumab combination as neoadjuvant treatment in localized stage III resectable cutaneous or mucosal melanoma patients.

Baseline and on-treatment PORTRAIT profiling, as described in the NEOREM Master Protocol (NCT07262489), will be performed using fresh blood and tumor samples. This profiling will reveal the immune status of patients and support biomarker-driven preselection for future trials.

DETAILED DESCRIPTION:
The combination of ipilimumab + nivolumab injected intravenously before resection of resectable stage III melanoma is more effective than adjuvant immunotherapy as recently demonstrated in a large phase III randomized controlled trial. However, the dual systemic immunotherapy gives rise to severe AEs (30% of patients had > grade 3 related AEs versus 14% in the adjuvant arm). NEO-1, a prospective, multicenter, phase II sub-protocol of the NEOREM master protocol (NCT07262489) focuses on evaluating the efficacy and safety of intratumoral neo-adjuvant treatment with ipilimumab and nivolumab in patients with resectable stage III melanoma.

NEO-1 is a proof-of-concept study designed to validate human intratumoral immunotherapy (HIT-IT) approach, which could maximize its dose/efficacy ratio of combined ipilimumab and nivolumab treatment while preventing systemic AEs. Image guided drug administration directly into tumor will increase the drug concentration at the tumor site leading to targeted drug action.

While evaluating the efficacy of intratumoral administration of ipilimumab in combination with nivolumab in melanoma patients, the NEO-1 study employs PORTRAIT profiling to analyze fresh blood and tumor samples collected at baseline and throughout treatment. This approach will reveal the features of the tumor microenvironment both before and after surgery, facilitating the identification of biomarkers that predict the efficacy of the proposed immunotherapy. The NEOREM master protocol (NCT07262489) allows the rapid analyses of the fresh samples collected, which enables an actual characterization of the immune landscape in patients prior to and during treatment.

ELIGIBILITY:
In addition to NEOREM Master Protocol inclusion and exclusion criteria, the following inclusion and exclusion criteria must be verified before inclusion in the NEO-1 trial:

Inclusion Criteria:

1. Patients ≥ 18 years old.
2. Patients with resectable and measurable (according to RECIST v1.1 criteria) stage III cutaneous and mucosal melanoma.
3. Patients who received anti-PD-1 and stopped treatment > 6 months prior to their inclusion in NEO-1 trial are eligible.
4. Patients who received target therapy and stopped treatment > 3 months prior to their inclusion in NEO-1 trial are eligible.

Exclusion Criteria:

1. Patients with clinically or radiologically detectable distant metastases.
2. Patients with uveal melanoma.
3. Patients with any hypersensitivity to the active ingredient or to any of the excipients of nivolumab and/ ipilimumab.
4. Patients without pathological evaluable disease according to RECIST v1.1 criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the efficacy of the intratumoral combination of ipilimumab and nivolumab in terms of pCR or MPR in patients with resectable stage III cutaneous or mucosal melanoma. | Between 6 and 8 weeks upon end of the treatment
  The primary efficacy endpoint is defined as a pathological complete response (pCR) rate defined as the percentage of patients with pCR defined as the complete absence of viable tumor cells, or the major pathologic response (MPR) defined as less than 10% of surviving tumor cells in tumor biopsy of the surgical specimen.
The primary objective is to evaluate the tolerability of the intratumoral combination of ipilimumab and nivolumab in patients with resectable stage III cutaneous or mucosal melanoma. | Between 6 and 8 weeks upon end of the treatment
  The primary safety endpoint defined as the percentage of patients whose surgery was delayed by more than 2 weeks beyond the planned timeline, due to treatment-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France